CLINICAL TRIAL: NCT06696443
Title: A Phase 3, Open-label Study Evaluating the Long-term Safety and Effectiveness of Suzetrigine in Subjects With Pain Associated With Diabetic Peripheral Neuropathy
Brief Title: Evaluation of the Long-term Safety and Effectiveness of Suzetrigine (SUZ) in Participants With Painful Diabetic Peripheral Neuropathy (DPN)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-548-112
Record Dates: First submitted 2024-11-15; First posted 2024-11-20 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Diabetic Peripheral Neuropathic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Suzetrigine (SUZ) (Experimental): Participants will receive SUZ once daily (qd) up to 52 weeks.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Tablets for oral administration.
  Other Names: VX-548; SUZ

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of SUZ and long-term effectiveness of SUZ in treating pain associated with DPN.

ELIGIBILITY:
Key Inclusion Criteria:

• Completed the final visit in the Treatment Period (i.e., Week 12) and subsequent 7-day period (to allow for taper of blinded capsule study drug) in a parent study such as VX24-548-110 or VX24-548-111

Key Exclusion Criteria:

* Any sensory abnormality (excluding DPN)
* History of drug intolerance in a parent study that would pose an additional risk to the participant in the opinion of the investigator
* Current participation in an investigational drug trial (other than a parent study)

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline up to Week 54

SECONDARY OUTCOMES:
Change From Baseline in Study 36-item Short-form Health Status (SF-36v2) Physical Component Summary (PCS) Score | From Baseline up to Week 52
Change From Baseline in the Short form McGill Pain Questionnaire-2 (SF-MPQ-2) Total Score | From Baseline up to Week 52

CONTACTS AND LOCATIONS:
Locations (65):
- United States (65):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - AMR Daphne, AL, Daphne, Alabama
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Neuro-Pain Medical Center, Fresno, California
  - Long Beach Research Institute, Long Beach, California
  - Angel City Research, Inc, Los Angeles, California
  - Empire Clinical Research, Pomona, California
  - Clinical Trials Research, Sacramento, California
  - Velocity Clinical Research, San Bernardino, San Bernardino, California
  - SCLA Management - Pain Management and Injury Relief, Thousand Oaks, California
  - Velocity Clinical Research - Denver, Englewood, Colorado
  - Velocity Clinical Research - Washington DC, Washington D.C., District of Columbia
  - AMR-Miami, Coral Gables, Florida
  - Accel Research - Deland, DeLand, Florida
  - Suncoast Research Associates - Miami, Doral, Florida
  - AMR Fort Myers (The Clinical Study Center), Fort Myers, Florida
  - Velocity Clinical Research - Hallandale Beach, Hallandale, Florida
  - CNS Healthcare - Jacksonville, Jacksonville, Florida
  - Accel Research Site - St. Petersburg/Largo, Largo, Florida
  - Accel Research Sites - Maitland, Maitland, Florida
  - 3Sync Research - Miami Lakes, Miami Lakes, Florida
  - Suncoast Clinical Research - New Port Richey, New Port Richey, Florida
  - Conquest Clinical Research - Orlando - Neuro, Orlando, Florida
  - Conquest Clinical Research - Winter Park, Winter Park, Florida
  - Accel Research - Decatur, Decatur, Georgia
  - Velocity Clinical Research - Boise, Meridian, Idaho
  - Feinberg School of Medicine - Anesthesiology, Chicago, Illinois
  - Healthcare Research Network - Flossmoor IL, Tinley Park, Illinois
  - Synexus Clinical Research - Evansville, Evansville, Indiana
  - AMR Wichita East, KS (Heartland Research Associates), Wichita, Kansas
  - AMR Lexington, Lexington, Kentucky
  - Velocity Clinical Research - Baton Rouge, Baton Rouge, Louisiana
  - Tandem Clinical Research- Covington, Covington, Louisiana
  - Mass General Brigham - Brigham and Women's Hospital - Main Campus, Boston, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Healthcare Research Network - Hazelwood MO, Hazelwood, Missouri
  - AMR Kansas City, Kansas City, Missouri
  - Velocity Clinical Research - Norfolk, Norfolk, Nebraska
  - HRI - Hassman Research Institute, Marlton, New Jersey
  - Velocity Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Swift Clinical OpCo, Inc, Brooklyn, New York
  - Velocity Clinical Research - Syracuse, East Syracuse, New York
  - Synexus Clinical Research - New York (DRS), New York, New York
  - Columbia Presbyterian - The Neurological Institute of New York, New York, New York
  - West Clinical Research, Morehead City, North Carolina
  - Eximia Research - Raleigh, Raleigh, North Carolina
  - Carolinas Pain Institute - Winston-Salem Office, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - Synexus Clinical Research - Cincinnati, Cincinnati, Ohio
  - META Medical Research Institute, Dayton, Ohio
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Suburban Research Associates - Media, Media, Pennsylvania
  - Velocity Clinical Research - Providence, East Greenwich, Rhode Island
  - Synexus Clinical Research- Anderson, Anderson, South Carolina
  - Clinical Trials of South Carolina - Charleston, Charleston, South Carolina
  - M3 Wake Research - Charleston, Charleston, South Carolina
  - Velocity Clinical Research - Spartanburg, Spartanburg, South Carolina
  - Zenos Clinical Research, Dallas, Texas
  - Be Well Clinical Studies - Austin, Round Rock, Texas
  - San Antonio Clinical Trials, San Antonio, Texas
  - Velocity Clinical Research - Waco, Waco, Texas
  - Kalo Clinical Research - Salt Lake City, Salt Lake City, Utah
  - Velocity Clinical Research - Salt Lake City, West Jordan, Utah
  - Dominion Medical Associates, Inc., Richmond, Virginia
  - Northwest Clinical Research Center (NWCRC), Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Siddiqui A, Xu JL, Abramowicz AE. Suzetrigine for the Treatment of Acute Pain: Comment. Anesthesiology. 2026 Feb 1;144(2):495-496. doi: 10.1097/ALN.0000000000005822. Epub 2025 Dec 11. No abstract available. PMID 41384808